CLINICAL TRIAL: NCT05672290
Title: Comparison of the Effects of External Electrical Stimulation Protocols in Women With Overactive Bladder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/01/03
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 will be applied external electric stimulation three days per week
  Interventions: Other: Electrical stimulation 1
- Group 2 (Active Comparator): Group 2 will be applied external electric stimulation one day per week
  Interventions: Other: Electrical stimulation 2

INTERVENTIONS:
Other: Electrical stimulation 1 — External electrical stimulation will be applied for 30 minutes 3 days a week during 6 weeks. Electrodes were placed around the pelvis.
  Arms: Group 1
Other: Electrical stimulation 2 — External electrical stimulation will be applied for 30 minutes one day a week during 6 weeks. Electrodes were placed around the pelvis.
  Arms: Group 2

SUMMARY:
The aim of our study is a comparison of the effects of external electrical stimulation protocols in women with overactive bladder (OAB).

DETAILED DESCRIPTION:
OAB is a condition defined by the International Continence Society as the presence of urinary urgency, usually accompanied by frequency and nocturia, with or without urgency urinary incontinence, in the absence of urinary tract infection or other obvious pathology. External electrical stimulation has positive effects on OAB. However, there are not enough studies on how often this stimulation is applied. Studies are needed on this subject.

ELIGIBILITY:
Inclusion Criteria:

* Being in the age range of 18-65 ,
* Having diagnosed with OAB,
* Being a volunteer

Exclusion Criteria:

* Being pregnant,
* presence of severe pelvic organ prolapse,
* malignant disease,
* urinary infection,
* neurological disease,
* have electronic and metal implant,
* loss of sensation,
* lumbosacral peripheral nerve lesion

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with overactive bladder
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Overactive bladder symptoms | change from baseline at 3 weeks and 6 weeks
  Overactive bladder symptoms will be assessed with the Overactive Bladder-V8 Questionnaire

SECONDARY OUTCOMES:
Urgency severity | change from baseline at 3 weeks and 6 weeks
  Urgency severity will be assessed with Patients' Perception of Intensity of Urgency Scale
Bladder functions | change from baseline at 3 weeks and 6 weeks
  Bladder functions will be assessed with voiding diary
Life quality | change from baseline at 3 weeks and 6 weeks
  Life quality will be assessed with the King's Health Questionnaire
Strength of pelvic floor muscle | change from baseline at 3 weeks and 6 weeks
  Strength of pelvic floor muscle will be assessed with Modified Oxford Scale
Perception of recovery | change from baseline at 3 weeks and 6 weeks
  Perception of recovery will be assessed with a 4-point Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University